CLINICAL TRIAL: NCT03183752
Title: The Role of Insulin Resistance and the Effect of Metformin Use on Volume of Benign Thyroid Nodules
Brief Title: Insulin Resistance and Metformin Use on Volume of Benign Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitário Clementino Fraga Filho (Other)
Responsible Party: Principal Investigator, Patricia Borges dos Santos, Principal Investigator, Hospital Universitário Clementino Fraga Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRUPO RINT
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Thyroid Nodule; Insulin Resistance
Keywords: thyroid; insulin; thyroid nodule; insulin resistance; thyroid volume; metformin
MeSH Terms: conditions — Thyroid Nodule; Insulin Resistance; Thyroid Diseases | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial with two groups: to use placebo or Metformine
Who Masked: Participant, Outcomes Assessor
Masking Description: The same researcher blinded regarding location group will access thyroid volume and thyroid nodule volume by ultrasound, in the beginning, six months and one year after randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): patients randomized to Metformin group
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): patients randomized to placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — 500 mg metformin three times daily
  Other Names: MTF
  Arms: Metformin
Drug: Placebo — 500 mg placebo three times daily
  Other Names: PLC
  Arms: Placebo

SUMMARY:
It has been shown that insulin might be involved in the pathogenesis of thyroid growth.

Objective To evaluate the impact of IR and metformin use on the volume of benign thyroid nodules (TNs).

Methods A randomized clinical trial to placebo (P) or MTF use. Previous fine needle aspiration confirming the diagnosis is necessary to inclusion. Patients will receive similar tablets of MTF and placebo and instruct to take 3 tablets/day of MTF (500mg/tablet). Thyroid volume, as TN volume, will be assess by ultrasound, both in the beginning, six months and one year after randomization, by the same researcher blinded regarding location group. Blood samples to measure: TSH, FT4, TPO-Ab, lipid profile, glucose and insulin were done after 8h fasting.

DETAILED DESCRIPTION:
It has been shown that insulin might be involved in the pathogenesis of thyroid growth. Previous studies suggest that metformin (MTF) therapy decreased thyroid volume and nodule size in subjects with insulin resistance (IR).

Objectives To evaluate the impact of IR and metformin use on the volume of benign thyroid nodules (TNs).

Methods A randomized clinical trial to placebo (P) or MTF use. Previous fine needle aspiration confirming the diagnosis is necessary to inclusion. Exclusion criteria were: nodules with a predominantly cystic pattern, pregnancy, diabetes, acromegaly, previous use of MTF, levothyroxine, corticoid or any weight loss medication in the past six months, hepatic or cardiac insufficiency, creatinine levels > 1.4 mg/dL and MTF intolerance doses >1.0 gram/day. Patients will receive similar tablets of MTF and placebo and will be instructed to take 3 tablets/day of MTF (500mg/tablet). Thyroid volume, as TN volume, will be accessed by ultrasound, both in the beginning, six months and one year after randomization, by the same researcher blinded regarding location group. Blood samples to measure: TSH, FT4, TPO-Ab, lipid profile, glucose and insulin were done after 8h fasting.

ELIGIBILITY:
Inclusion Criteria:

* patients with benign nodules diagnosed by fine needle aspiration biopsy (FNAB)

Exclusion Criteria:

* Nodules with a predominantly cystic pattern
* Eggshell calcification
* Coalescent thyroid nodules (not suitable for size analysis)
* Pregnancy
* Diabetes
* Acromegaly
* Previous use of MTF, levothyroxine, corticoid or any weight loss medication in the past six months
* Hepatic or cardiac insufficiency
* Creatinine levels > 1.4 mg/dL
* MTF intolerance doses < 1.0 gram/day

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-08-13; Primary Completion 2018-10-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
changes in nodule volume from baseline after metformin use | one year
  the impact of metformin on the volume of thyroid nodules

SECONDARY OUTCOMES:
changes in nodule volume from baseline and changes in homa-ir | one year
  the impact of insulin resistance in volume of thyroid nodules
changes in TSH levels from baseline after metformin use | one year
  the impact of metformin use in TSH levels

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Santos, MD, Principal Investigator — UFRJ; Patricia Teixeira, PhD, Study Director — UFRJ
Locations (1):
- Patricia Santos, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No